CLINICAL TRIAL: NCT05261698
Title: Effects of Routine Physical Therapy With and Without Home-Based Exercise Manual on Pain and Disability in Patients of Postural Neck Pain: A Randomized Clinical Trial
Brief Title: Effects of Home-Based Exercise Manual on Pain and Disability in Patients of Postural Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ULahore Muhammad Adil
Record Dates: First submitted 2022-02-19; First posted 2022-03-02 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Postural Neck Pain
Keywords: Postural Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arms (Active Comparator): Control group: in control group moist heating pads along with TENS shall be applied on neck for 10 minutes and then neck isometrics and strengthening exercises shall be performed.
  Interventions: Other: Conventional PT
- Assigned Interventions (Experimental): Experimental group: in the experimental group we will provide moist heating pads along with TENS on the neck for 10 minutes and then neck isometrics and strengthening exercises shall be performed. Patients in the experimental group will also receive a home-based exercise manual.
  Interventions: Other: Home-based Exercise Manual

INTERVENTIONS:
Other: Home-based Exercise Manual — in the experimental group we will provide moist heating pads along with TENS on the neck for 10 minutes and then neck isometrics and strengthening exercises shall be performed. Patients in the experimental group will also receive a home-based exercise manual.
  Arms: Assigned Interventions
Other: Conventional PT — In this group patients will receive routine physical therapy including hot pack for 10 minutes, stretching, strengthening exercise and TENS at the end of each session.
  Arms: Arms

SUMMARY:
The main aim of this study is to determine the effects of routine physical therapy with and without home-based exercise manual on pain and disability in patients of postural neck pain. To exceptional time, the effects and outcomes of home-based exercise manual for the patients with postural neck pain have not yet been explored. Due to the current Covid-19 pandemic and social isolation, most of the individuals with office based occupations are performing their duties from their homes, which has some negative impact on their neck biomechanics and leads to the postural neck pain, this study will not only enlighten the beneficial effects of home-based exercise manual for the patients of postural neck pain, to reduce the risk of disability and improve their quality of life, but it will also be cost effective for them.

DETAILED DESCRIPTION:
After back pain, most commonly found musculoskeletal ailment is the neck pain. Due to the poor neck posture, postural neck pain appears. It is estimated that, about 60% of the neck pain patients' have the forward head posture. Many people visit hospitals or other medical centers at least once in their life due to this problem.

Those individuals with chronic neck pain who work in offices, industries or perform other computer-based tasks, that require sitting for longer period of time have altered postural behaviors. Persistent neck pain has the negative impact as it has the potential to change the biomechanics of cervical spine specifically in individuals who spend most of their time in sitting position in front of computer screens. Continuous postural neck pain may lead to the forward head posture that rises load on the posterior structures of the cervical spine such as ligaments, muscles, bones and joint capsules and brings changes in scapular kinetics and kinematics.

According to the previous researches, forward head posture causes tightening of the shoulder and anterior neck muscles, shortening of the posterior neck extensors, and affects the kinematics and position of the scapula. Proper posture of the body is believed to be the state in which there is a musculoskeletal balance and minimal amount of strain and stress on the body. However most of the people are not able to maintain that equilibrium in the musculoskeletal structures of the body.

An ideal posture is considered only when the external auditory meatus is lined up with the vertical postural line. As seen in in the lateral view, the vertical line passes through external auditory meatus, the shoulder joint, slightly behind the hip joint, through the center of the knee joint and slightly in front of the ankle joint. Postural neck pain is believed to be associated with the forward head posture and is one of the common types of poor head posture seen in patients with neck disorders.

Neck pain is the most commonly occurring clinical condition, and its associated social and economic costs related to disability and days off work are just about equal to the lumbar pain. Individuals with the postural neck pain have been reported with the change in muscular control such as increased activity of the superficial muscles of the cervical spine and upper trapezius. Although the exact association between posture and neck pain is unresolved. Cervical neck posture is believed to have impact on dorsal neck muscle activity during lifting or even at rest. Moreover, postural neck pain may lead to the forward head posture linked with the thoracic kyphosis which has indirect impact on the rotational range of motion and cervical flexion. Occupations with sustained computer use and prolong computer usage may lead to the functional kyphosis, that seems to affect posture of the neck and scapular positioning and activity of the upper trapezius. Modifications in the workplace environment and postural correction have been shown in reducing postural neck pain.

The main aim of the study is to compare the effects of routine physical therapy with and without home-based exercise manual on pain and disability in patients of postural neck pain.

ELIGIBILITY:
Inclusion Criteria:

* All patients with postural neck pain aged 18-60 years shall be included.
* Patients experiencing postural neck pain at least once a week.
* A symptom duration of greater than 3 months.
* Postural neck pain that is aggravated by the sustained postural loading, and relieved by postural modification.
* Patients who are able to read and write.

Exclusion Criteria:

* Neck pain due to specific causes i.e. disc protrusion, radicular syndrome
* Any accidental injury of spine
* Inflammatory rheumatic disease
* Congenital deformity of the spine
* Spinal canal stenosis
* Neoplasm
* Females who are pregnant
* Patients who had spinal surgery within the previous 12 months or any other invasive treatment of the spine within the previous 4 weeks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | 2 weeks
  Pain will be measured by Numerical Pain Rating Scale (NPRS), in which patients are asked to circle the number between 0 and 10. The numerical scale is most commonly 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable." The patient picks (verbal version) or draws a circle around.
Neck Disability Index (NDI) | 2 weeks
  The Neck Disability Index (NDI) is a self-report questionnaire which is used to determine how neck pain affects a patient's daily life and to assess the self-rated disability of patients with neck pain. This questionnaire is used to gather the details about the intensity of neck pain among patients that has affected the capability to manage in daily routine. Every single section of this questionnaire is scored on a 0 to 5 rating scale, in which 0 means "no pain" whereas 5 means "worst imaginable pain".

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Adil, MPHIL-MSK*, Principal Investigator — University of Lahore
Locations (1):
- Pakistan Society for Rehabilitation of the Disabled, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta BD, Aggarwal S, Gupta B, Gupta M, Gupta N. Effect of Deep Cervical Flexor Training vs. Conventional Isometric Training on Forward Head Posture, Pain, Neck Disability Index In Dentists Suffering from Chronic Neck Pain. J Clin Diagn Res. 2013 Oct;7(10):2261-4. doi: 10.7860/JCDR/2013/6072.3487. Epub 2013 Oct 5. PMID 24298492
- [Background] Argent R, Daly A, Caulfield B. Patient Involvement With Home-Based Exercise Programs: Can Connected Health Interventions Influence Adherence? JMIR Mhealth Uhealth. 2018 Mar 1;6(3):e47. doi: 10.2196/mhealth.8518. PMID 29496655
- [Background] Cramer H, Lauche R, Hohmann C, Ludtke R, Haller H, Michalsen A, Langhorst J, Dobos G. Randomized-controlled trial comparing yoga and home-based exercise for chronic neck pain. Clin J Pain. 2013 Mar;29(3):216-23. doi: 10.1097/AJP.0b013e318251026c. PMID 23249655
- [Background] Fakhry F, Spronk S, de Ridder M, den Hoed PT, Hunink MG. Long-term effects of structured home-based exercise program on functional capacity and quality of life in patients with intermittent claudication. Arch Phys Med Rehabil. 2011 Jul;92(7):1066-73. doi: 10.1016/j.apmr.2011.02.007. PMID 21704786
- [Background] Baggetta R, D'Arrigo G, Torino C, ElHafeez SA, Manfredini F, Mallamaci F, Zoccali C, Tripepi G; EXCITE Working group. Effect of a home based, low intensity, physical exercise program in older adults dialysis patients: a secondary analysis of the EXCITE trial. BMC Geriatr. 2018 Oct 20;18(1):248. doi: 10.1186/s12877-018-0938-5. PMID 30342464
- [Background] Damasceno GM, Ferreira AS, Nogueira LAC, Reis FJJ, Andrade ICS, Meziat-Filho N. Text neck and neck pain in 18-21-year-old young adults. Eur Spine J. 2018 Jun;27(6):1249-1254. doi: 10.1007/s00586-017-5444-5. Epub 2018 Jan 6. PMID 29306972
- [Background] Korakakis V, O'Sullivan K, O'Sullivan PB, Evagelinou V, Sotiralis Y, Sideris A, Sakellariou K, Karanasios S, Giakas G. Physiotherapist perceptions of optimal sitting and standing posture. Musculoskelet Sci Pract. 2019 Feb;39:24-31. doi: 10.1016/j.msksp.2018.11.004. Epub 2018 Nov 17. PMID 30469124
- [Background] Im B, Kim Y, Chung Y, Hwang S. Effects of scapular stabilization exercise on neck posture and muscle activation in individuals with neck pain and forward head posture. J Phys Ther Sci. 2016 Mar;28(3):951-5. doi: 10.1589/jpts.28.951. Epub 2016 Mar 31. PMID 27134391
- [Background] Edmondston S, Bjornsdottir G, Palsson T, Solgard H, Ussing K, Allison G. Endurance and fatigue characteristics of the neck flexor and extensor muscles during isometric tests in patients with postural neck pain. Man Ther. 2011 Aug;16(4):332-8. doi: 10.1016/j.math.2010.12.005. Epub 2011 Jan 20. PMID 21256071
- [Background] Mani S, Sharma S, Singh DK. Concurrent validity and reliability of telerehabilitation-based physiotherapy assessment of cervical spine in adults with non-specific neck pain. J Telemed Telecare. 2021 Feb;27(2):88-97. doi: 10.1177/1357633X19861802. Epub 2019 Jul 4. PMID 31272309
- [Background] Nasir MF, Jawed R, Baig NN, Younus M, Arshad A, Tahir A. A study to observe the effects of physiotherapy with and without manual therapy in the management postural neck pain: A randomized control trial. J Pak Med Assoc. 2021 Jan;71(1(A)):8-11. doi: 10.47391/JPMA.186. PMID 33484509
- [Background] Wegner S, Jull G, O'Leary S, Johnston V. The effect of a scapular postural correction strategy on trapezius activity in patients with neck pain. Man Ther. 2010 Dec;15(6):562-6. doi: 10.1016/j.math.2010.06.006. Epub 2010 Jul 21. PMID 20663706
- [Background] Pillastrini P, de Lima E Sa Resende F, Banchelli F, Burioli A, Di Ciaccio E, Guccione AA, Villafane JH, Vanti C. Effectiveness of Global Postural Re-education in Patients With Chronic Nonspecific Neck Pain: Randomized Controlled Trial. Phys Ther. 2016 Sep;96(9):1408-16. doi: 10.2522/ptj.20150501. Epub 2016 Mar 24. PMID 27013576
- [Background] Richards KV, Beales DJ, Smith AJ, O'Sullivan PB, Straker LM. Neck Posture Clusters and Their Association With Biopsychosocial Factors and Neck Pain in Australian Adolescents. Phys Ther. 2016 Oct;96(10):1576-1587. doi: 10.2522/ptj.20150660. Epub 2016 May 12. PMID 27174256